CLINICAL TRIAL: NCT04286529
Title: Effect of 1,25-dihydroxyvitamin D3, Treatment on Insulin Secretion and Muscle Strength in Pre-diabetic Persons
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty with study logistics due to COVID-19
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rajiv Kumar, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-010890
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Results first posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-02

CONDITIONS: Pre-Diabetic
Keywords: Pre-menopausal women
MeSH Terms: conditions — Glucose Intolerance | interventions — Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Men-Calcitriol (Active Comparator): Calcitriol (1,25(OH)2D3) 0.25mcg capsule daily for eight weeks.
  Interventions: Drug: Calcitriol capsules
- Premenopausal Women-Calcitriol (Active Comparator): Calcitriol (1,25(OH)2D3) 0.25mcg capsule daily for eight weeks.
  Interventions: Drug: Calcitriol capsules
- Men-Placebo (Placebo Comparator): 0.25mcg capsule daily for eight weeks
  Interventions: Drug: Oral Placebo
- Premenopausal Women-Placebo (Placebo Comparator): 0.25mcg capsule daily for eight weeks
  Interventions: Drug: Oral Placebo

INTERVENTIONS:
Drug: Calcitriol capsules — 0.25micrograms, taken daily for eight weeks, orally
  Arms: Men-Calcitriol; Premenopausal Women-Calcitriol
Drug: Oral Placebo — Placebo will be created to mimic the appearance of the study drug
  Arms: Men-Placebo; Premenopausal Women-Placebo

SUMMARY:
The purpose of this research is to study the effects of 1,25(OH)2 D3 (a prescription form of active Vitamin D) on muscle strength and insulin secretion by the pancreas and glucose utilization by skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of >24kg/m2
* Fasting serum glucose <126 mg/dL

Exclusion Criteria:

* BMI</=24 kg/m2
* Fasting serum glucose >/=126 mg/dL
* Patient is taking Calcium or Vitamin D supplements and is unwilling to stop for 8 weeks
* Serum Calcium >10.2 mg/dL
* Serum inorganic phosphorous >4.5mg/dL
* Pregnancy or breastfeeding
* Diagnosis of Diabetes Mellitus
* Diagnosis of Rheumatoid Arthritis
* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Renal in sufficiency/failure ( serum creatinine >1.5 mg/dL men, > 1.3 mg/dL women)
* Chronic active liver disease (bilirubin >1.2 mg/dL, AST>144IU/L, or ALT >165 IU/L)
* History of chronic hepatitis
* Active coronary artery disease ( unstable angina, myocardial infarction, stroke and revascularization of coronary, peripheral or carotid artery within the last 3 months)
* Oral warfarin group medications or history of blood clotting disorders
* Platelet count <100,000 per uL within the last 7 days
* Alcohol consumption greater than 2 glasses/day or other substance abuse
* Untreated or uncontrolled thyroid disorders (outside a TSH range of 0.5 to 10mIU/L)
* Debilitating chronic disease (at the discretion of the investigators)
* The presence of infections, highly communicable diseases ( AIDS, active tuberculosis, venereal disease, hepatitis)
* Any malignancy

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menopausal status is of interest to the study.
Enrollment: 17 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajiv Kumar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
Started | 4 | 4 | 5 | 4
Completed | 3 | 1 | 3 | 1
Not Completed | 1 | 3 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo | Total
Number analyzed (Participants) | 4 | 4 | 5 | 4 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (4.2) | 29 (5.2) | 30 (2.6) | 27 (2.6) | 30 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 0 | 4 | 8
  Male | 4 | 0 | 5 | 0 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 4 | 3 | 4 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Glucose Levels
Description: Blood will be obtained to measure glucose after a glucose tolerance test. The glucose tolerance test involves an overnight fast and then participants will ingest a drink containing 75 grams of glucose with blood obtained over a 120 minute period.
Time Frame: Baseline and 8 weeks
Population: Data not collected or analyzed at 8 weeks for the one participant in the Premenopausal Women-Placebo study arm.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
Number analyzed (Participants) | 3 | 1 | 3 | 1
mg/dL
  Baseline | 90 (4.1) | 76 (0) | 89 (4) | 82 (0)
  8 weeks: number analyzed (Participants) | 3 | 1 | 3 | 0
  8 weeks | 98 (9.2) | 85 (0) | 85 (4.7) |

2. Primary Outcome: Insulin Level
Description: Blood will be obtained to measure insulin level after a glucose tolerance test. The glucose tolerance test involves an overnight fast and then participants will ingest a drink containing 75 grams of glucose with blood obtained over a 120 minute period.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: uIU/mL
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
Number analyzed (Participants) | 3 | 1 | 3 | 1
uIU/mL
  Baseline | 4.7 (1.8) | 4.6 (0) | 3 (1.6) | 2.4 (0)
  8 Weeks | 5 (1.8) | 4 (0) | 3 (0.8) | 4 (0)

3. Primary Outcome: C-Peptide Level
Description: Blood will be obtained to measure c-peptide level after a glucose tolerance test. The glucose tolerance test involves an overnight fast and then participants will ingest a drink containing 75 grams of glucose with blood obtained over a 120 minute period.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
Number analyzed (Participants) | 3 | 1 | 3 | 1
nmol/L
  Baseline | 0.6 (0.07) | 0.5 (0) | 0.7 (0.3) | 0.5 (0)
  8 Weeks | 0.74 (0.07) | 0.55 (0) | 0.49 (0.08) | 0.52 (0)

4. Secondary Outcome: PROMIS 10 Questionnaire
Description: Brief 10 question multiple choice survey
Time Frame: 8 weeks
Population: Data not collected or analyzed
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 9 weeks on all participants.
Arm/Group | Men-Calcitriol | Premenopausal Women-Calcitriol | Men-Placebo | Premenopausal Women-Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 0/5 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Men-Calcitriol (N=4) | Premenopausal Women-Calcitriol (N=4) | Men-Placebo (N=5) | Premenopausal Women-Placebo (N=4)
Deep ache medial and lateral parapatellar region (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2000-03-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04286529/Prot_SAP_000.pdf